CLINICAL TRIAL: NCT03867201
Title: A 12-week Phase 3, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Once Monthly Subcutaneous Erenumab 70 mg in Adult Chronic Migraine Patients
Brief Title: Study of Efficacy and Safety of Erenumab in Adult Chronic Migraine Patients
Acronym: DRAGON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAMG334A2304
Record Dates: First submitted 2019-02-25; First posted 2019-03-07 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: AMG334; erenumab; migraine; chronic; headache; Chinese
MeSH Terms: conditions — Migraine Disorders; Bronchiolitis Obliterans Syndrome; Headache | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erenumab (Experimental): Administered by pre-filled syringe
  Interventions: Biological: Erenumab
- Placebo (Placebo Comparator): Administered by pre-filled syringe
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Erenumab — Administered by pre-filled syringe
  Other Names: AMG334
  Arms: Erenumab
Other: Placebo — Administered by pre-filled syringe
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of erenumab in patients with chronic migraine in Asian population.

DETAILED DESCRIPTION:
This study used a single-cohort, 2-treatment arms, randomized (1:1 (70 mg:placebo)), double-blind study design in adult subjects with chronic migraine. A screening period of 2 weeks was used to assess initial eligibility, followed by a 4-week baseline period to assess diary compliance and headache frequency.

Eligible patients were then randomized to either erenumab 70 mg or placebo for 12 weeks, followed by an open-label treatment period to last until end of PTA determined by the product launch in the country or the country's decision not to launch. A safety follow-up visit occurred 12 weeks after the last treatment for subjects who discontinue the double-blind treatment or who completed the double-blind treatment period without continuing in the open-label treatment period.

ELIGIBILITY:
key inclusion Criteria:

1. History of at least 5 attacks of migraine
2. ≥ 15 headache days of which ≥ 8 headache days meet criteria as migraine days during the baseline period
3. >=80% diary compliance during the baseline period

Key exclusion Criteria:

1. Older than 50 years of age at migraine onset
2. History of cluster or hemiplegic headache
3. Evidence of seizure or major psychiatric disorder
4. Cardiac or active hepatic disease
5. Pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- China (23):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Xiamen, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Jingzhou, Hubei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
- India (3):
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
- Malaysia (4):
  - Novartis Investigative Site, Seberang Jaya, Pulau Pinang
  - Novartis Investigative Site, Sungai Buloh, Selangor
  - Novartis Investigative Site, Kuala Terengganu, Terengganu
  - Novartis Investigative Site, Kuala Lumpur
- Philippines (2):
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Pasig
- Novartis Investigative Site, Singapore, Singapore
- South Korea (4):
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Taiwan (6):
  - Novartis Investigative Site, Chiayi City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taichung County
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (4):
  - Novartis Investigative Site, Bangkok, THA
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Vietnam (2):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Yu S, Kim BK, Wang H, Zhou J, Wan Q, Yu T, Lian Y, Arkuszewski M, Ecochard L, Wen S, Yin F, Li Z, Su W, Wang SJ. A phase 3, randomised, placebo-controlled study of erenumab for the prevention of chronic migraine in patients from Asia: the DRAGON study. J Headache Pain. 2022 Nov 21;23(1):146. doi: 10.1186/s10194-022-01514-9. PMID 36404301
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2604

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A screening period of 2 weeks was used to assess initial eligibility, followed by a 4-week baseline period to assess diary compliance and headache frequency.
Groups:
- Erenumab 70 mg: Administered by pre-filled syringe every 4 weeks starting at Day 1
- Placebo: Placebo administered by pre-filled syringe at Day 1 and Weeks 4 and 8. Erenumab 70 mg administered by pre-filled syringe every 4 weeks starting at Week 12
Period: Double-Blind Period Until Week 12
Arm/Group | Erenumab 70 mg | Placebo
Started | 279 | 278
Completed | 273 | 272
Not Completed | 6 | 6
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Pregnancy | 1 | 1
Not completed — Adverse Event | 2 | 1
Period: Open-Label Period From Week 12
Arm/Group | Erenumab 70 mg | Placebo
Started | 224 | 232
Completed | 105 | 121
Not Completed | 119 | 111
Not completed — Adverse Event | 5 | 11
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 6 | 3
Not completed — Pregnancy | 2 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 90 | 85
Not completed — No longer clinically benefiting | 12 | 10
Not completed — New Therapy for Study Indication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Erenumab 70 mg; Placebo: Administered by pre-filled syringe at Day 1 and Weeks 4 and 8
- Total: Total of all reporting groups
Arm/Group | Erenumab 70 mg | Placebo | Total
Number analyzed (Participants) | 279 | 278 | 557
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (10.9) | 41.9 (10.9) | 41.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 237 | 454
  Male | 62 | 41 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 277 | 275 | 552
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days During the Last 4 Weeks of the 12-week Treatment Period
Description: A migraine day was defined as any calendar day in which the subject experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for ≥4 continuous hours, and meeting at least one of the following criteria:
  1. ≥2 of the following pain features:
     * Unilateral
     * Throbbing
     * Moderate to severe
     * Exacerbated with exercise/physical activity
  2. ≥1 of the following associated symptoms:
     * Nausea and/or vomiting
     * Photophobia and phonophobia
Time Frame: baseline (4 weeks period prior to start of study drug), week 9 to 12
Population: Full Analysis Set. All randomized participants with evaluable measurements at the respective timepoint.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Erenumab 70 mg | Placebo
Number analyzed (Participants) | 270 | 274
days | -8.19 (0.46) | -6.62 (0.45)
Statistical Analysis 1: Comparison: Erenumab 70 mg vs Placebo; Test type: Superiority; p = 0.015, Mixed Models Analysis; Mean Difference (Net) = -1.57, 95% CI 2-sided [-2.83 to -0.30], Standard Error of Mean 0.64

2. Secondary Outcome: Change From Baseline in Migraine-related Disability and Productivity as Measured by the mMIDAS During the Last 4 Weeks of the 12-week Treatment Period
Description: The modified MIDAS is a 5-item self-administered questionnaire that sums the number of productive days lost over the past month in two settings: the workplace and the home. The MIDAS also assesses disability in family, social, and leisure activities. The MIDAS score is the sum of missed days due to a headache from paid work, housework, and non-work (family, social, leisure) activities; and days at paid work or housework where productivity was reduced by at least half.
Time Frame: baseline (4 weeks period prior to start of study drug), week 9 to 12
Population: Full Analysis Set. All randomized participants with evaluable measurements at the respective timepoint.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Erenumab 70 mg | Placebo
Number analyzed (Participants) | 263 | 268
days | -14.67 (1.20) | -12.93 (1.19)

3. Secondary Outcome: Number of Participants With at Least 50% Reduction From Baseline in Monthly Migraine Days During the Last 4 Weeks of the 12-week Treatment Period
Description: as for outcome 1
Time Frame: baseline (4 weeks period prior to start of study drug), week 9 to 12
Population: Full Analysis Set. All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab 70 mg | Placebo
Number analyzed (Participants) | 279 | 278
Participants | 131 | 102

4. Secondary Outcome: Change From Baseline in Monthly Acute Headache Medication Days During the Last 4 Weeks of the 12-week Treatment Period
Description: An acute headache medication day was defined as a day when medication was taken to treat acute headache.
Time Frame: baseline (4 weeks period prior to start of study drug), week 9 to 12
Population: Full Analysis Set. All randomized participants with evaluable measurements at the respective timepoint.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Erenumab 70 mg | Placebo
Number analyzed (Participants) | 270 | 274
days | -5.34 (0.39) | -4.66 (0.39)

5. Secondary Outcome: Number of Subjects With Adverse Events as a Measure of Safety
Description: Number of subjects with adverse events was assessed separately in the double-blind treatment period (DBTP) and the open-label treatment period (OLTP).
Time Frame: DBTP: 12 weeks for participants entering the OLTP. 20 weeks for participants NOT entering the OLTP. OLTP: From week 12 until up to approximately 4 years.
Population: Safety Set (for DBTP). Number of participants entering the OLTP (for OLTP).
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab 70 mg | Placebo
Number analyzed (Participants) | 279 | 278
Participants
  Double-Blind Treatment Period: Number of subjects with at least one AE | 127 | 132
  Open-Label Treatment Period: Number of subjects with at least one AE: number analyzed (Participants) | 224 | 232
  Open-Label Treatment Period: Number of subjects with at least one AE | 152 | 176

6. Secondary Outcome: Number of Subjects With Anti-AMG 334 Antibodies
Description: anti-AMG 334 antibodies assessed for binding and neutralizing)
Time Frame: baseline, 20 weeks
Population: FAS including participants with a valid assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab 70 mg | Placebo
Number analyzed (Participants) | 266 | 264
Participants
  Binding antibody positive at baseline: number analyzed (Participants) | 265 | 262
  Binding antibody positive at baseline | 0 | 0
  Neutralizing antibody positive at baseline: number analyzed (Participants) | 265 | 262
  Neutralizing antibody positive at baseline | 0 | 0
  Binding antibody positive at any time from baseline to week 20 | 9 | 0
  Neutralizing antibody positive at any time from baseline to week 20 | 1 | 0

ADVERSE EVENTS:
Time Frame: Double-Blind Treatment Period: 12 weeks for participants entering the open-label treatment period. 20 weeks for participants NOT entering the open-label treatment period. Open-Label Treatment Period: From week 12 until up to approximately 4 years.
Groups:
- Erenumab 70mg DBTP; Placebo DBTP: double-blind treatment period (DBTP). Administered by pre-filled syringe at Day 1 and Weeks 4 and 8.
- Erenumab 70mg OLTP (Erenumab 70mg in DBTP); Erenumab 70mg OLTP (Placebo in DBTP): open-label treatment period (OLTP). Administered by pre-filled syringe every 4 weeks starting at week 12.
Arm/Group | Erenumab 70mg DBTP | Placebo DBTP | Erenumab 70mg OLTP (Erenumab 70mg in DBTP) | Erenumab 70mg OLTP (Placebo in DBTP)
All-Cause Mortality (participants affected / at risk) | 0/279 | 0/278 | 0/224 | 0/232
Serious Adverse Events (participants affected / at risk) | 7/279 | 7/278 | 21/224 | 24/232
Other Adverse Events (participants affected / at risk) | 58/279 | 59/278 | 92/224 | 120/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab 70mg DBTP (N=279) | Placebo DBTP (N=278) | Erenumab 70mg OLTP (Erenumab 70mg in DBTP) (N=224) | Erenumab 70mg OLTP (Placebo in DBTP) (N=232)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 2 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hyperplasia adrenal (Endocrine disorders) | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 1
Cataract cortical (Eye disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Chronic hepatitis B (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint capsule rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Endometrial stromal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intraductal papillary breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 2 | 1
Cystitis glandularis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine adhesions (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab 70mg DBTP (N=279) | Placebo DBTP (N=278) | Erenumab 70mg OLTP (Erenumab 70mg in DBTP) (N=224) | Erenumab 70mg OLTP (Placebo in DBTP) (N=232)
Constipation (Gastrointestinal disorders) | 24 | 11 | 14 | 29
COVID-19 (Infections and infestations) | 0 | 1 | 39 | 47
Nasopharyngitis (Infections and infestations) | 10 | 5 | 6 | 13
Upper respiratory tract infection (Infections and infestations) | 16 | 19 | 31 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 12
Dizziness (Nervous system disorders) | 5 | 12 | 10 | 17
Headache (Nervous system disorders) | 1 | 6 | 13 | 12
Migraine (Nervous system disorders) | 4 | 6 | 3 | 15
Insomnia (Psychiatric disorders) | 4 | 5 | 9 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT03867201/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03867201/SAP_001.pdf